CLINICAL TRIAL: NCT06760494
Title: Prediction of Microvascular Invasion in HCC Using Spatiotemporal Radiomics of Contrast-enhanced Ultrasound: a Deep Learning Model With Transcriptomics Correlation
Brief Title: Microvascular Invasion Artificial Intelligence Prediction Via Contrast-enhanced Ultrasound With Explainability
Acronym: MAPUSE
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Other Study IDs: MAPUSE; 92159305 (Other: The National Natural Science Foundation of China); 82030047 (Other: The National Natural Science Foundation of China); 82325027 (Other: The National Natural Science Foundation of China)
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: HCC - Hepatocellular Carcinoma; Microvascular Invasion (MVI)
Keywords: hepatocellular carcinoma; microvascular invasion; contrast-enhanced ultrasound; deep learning
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chinese PLA General Hospital Cohort: Patients from Chinese PLA General Hospital (northern China) after surgical treatment
  Interventions: Diagnostic Test: the MAPUSE model
- the First Affiliated Hospital of Sun Yat-sen University Cohort: Patients from the First Affiliated Hospital of Sun Yat-sen University (southern China) after surgical treatment
  Interventions: Diagnostic Test: the MAPUSE model

INTERVENTIONS:
Diagnostic Test: the MAPUSE model — Using the MAPUSE model to predict MVI status before surgical resection for HCC patients

SUMMARY:
An artificial intelligence (AI) model to predict MVI of HCC using contrast-enhanced ultrasound was constructed. This model also has biological explainability. The investigators named it as MAPUSE (MVI AI prediction via contrast-enhanced ultrasound with explainability).

The goal of MAPUSE study is to prospectively test the performance of MAPUSE model on MVI prediction and its biological correlation in different geographical areas of China.

DETAILED DESCRIPTION:
The presence of microvascular invasion (MVI) in hepatocellular carcinoma (HCC) is a critical prognostic indicator, but its preoperative diagnosis remains challenging. Contrast-enhanced ultrasound (CEUS), with its dynamic microvascular imaging capability, holds promise in prediction of MVI.

The investigators constructed an artificial intelligence (AI) model to predict MVI using contrast-enhanced ultrasound. This model also has biological explainability. We named it as MAPUSE (MVI AI prediction via contrast-enhanced ultrasound with explainability).

The goal of MAPUSE study is to prospectively test the performance of MAPUSE model on MVI prediction and its biological correlation in different geographical areas of China.

The performance of MAPUSE is to be tested in two prospective testing cohorts from two centers in southern and northern China. Before surgery, patient CEUS videos will be collected and analysed by MAPUSE model to generate an MVI risk score. According to the postoperative pathological diagnosis of MVI (golden criterion), the result of MAPUSE will be evaluated. Parameters include area under curve (AUC), accuracy (ACC), sensitivity, specificity and F1-score.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. The HCC diagnosis and the presence of MVI were confirmed by surgical pathology.
3. Complete and clear CEUS videos obtained within two weeks preoperatively.

Exclusion Criteria:

1. Unqualified CEUS images.
2. Missing surgical pathological diagnosis.
3. Lesions underwent local treatments.
4. Non-HCC diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent surgical treatment for HCC
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
area under operating characteristic curves (AUC) | From preoperative enrollment to the postoperative confirmation of pathological diagnosis (7-15 days postopertively)
  the area under operating characteristic curves (AUC) to evaluate the performance of MAPUSE model in predicting MVI in HCC patients

SECONDARY OUTCOMES:
ACC (accuracy) | From preoperative enrollment to the postoperative confirmation of pathological diagnosis (7-15 days postopertively)
  The ratio of the number of samples correctly predicted by the model to the total number of samples
Specificity | From preoperative enrollment to the postoperative confirmation of pathological diagnosis (7-15 days postopertively)
  Proportion of all patients without MVI who are predicted negative by MAPUSE
Sensitivity | From preoperative enrollment to the postoperative confirmation of pathological diagnosis (7-15 days postopertively)
  The proportion of patients with MVI that MAPUSE correctly identifies

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Pang, Principal Investigator — Chinese PLA General Hospital
Locations (2):
- China (2):
  - the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided